CLINICAL TRIAL: NCT01251042
Title: A Prospective, Randomized, Controlled Study on Intra-operative Autologous Transfusion With the Sangvia® Blood Salvage System in Spinal Surgery
Brief Title: Comparison Between Return and Wastage of Your Own Blood, Collected During Spinal Surgery, for Verification of Safety When Returning Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-DRA-0006
Record Dates: First submitted 2010-09-24; First posted 2010-12-01 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2013-04

CONDITIONS: Spinal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sangvia and retransfusion (Experimental)
  Interventions: Device: Sangvia
- Sangvia and no retransfusion (Sham Comparator)
  Interventions: Device: Sangvia

INTERVENTIONS:
Device: Sangvia — The Sangvia® Blood Salvage System used to collect blood intra-operatively.

SUMMARY:
The study is an open, randomized, controlled, single-centre study including a total of 42 evaluable subjects scheduled for spinal surgery with an approximate expected bleeding of 800-1500 ml. The Sangvia® Blood Salvage System will be set up for all subjects to collect blood intra-operatively. When the transfusion bag is filled, i.e. when around 500 ml of blood has been collected, the subject will be randomized to either be retransfused with the blood collected (investigational group) or not (control group). The primary objective for this study is to investigate the blood quality and isolate the systemic effects in intra-operatively collected blood. The systemic p-Hb concentration has been chosen as the primary outcome variable based on previous experience and literature and is considered as the major safety concern for the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Male and female subjects aged 18 years and over subjected to spinal surgery with an approximate expected bleeding of 800-1500 ml.
* Subjects classified as ASA Physical Status Classification System class P1, P2 or P3 according to the American Society of Anaesthesiology.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site).
* Previous enrolment or randomisation of treatment in the present study.
* Participation in another clinical study, that may interfere with the present study.
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech.
* Haemophilia.
* Hyperkalemia (i.e. values above the normal reference values at study site).
* Symptoms of impaired renal function including creatinine clearance levels (using the Cockcroft-Gault formula) <30 ml/min.
* Malignancy in the area of the operative site.
* Current or expected use of cytotoxic drugs.
* Symptoms of systemic infection or local infection in the operation field.
* Pregnancy.
* Sickle cell anaemia and/or pre-operative Hb concentration <11 g/dl (6,8 mmol/l).
* Use of recombinant erythropoietin (EPO) or fibrin sealant.
* Use of other autologous blood transfusion than with the Sangvia® system (e.g. CellSaver and pre-donation) or other blood saving techniques (e.g. normovolemic hemodilution).
* Hypotensive anesthesia.
* Use of antithrombotic medication within 5 days of surgery (NSAID, Clopidogrel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rud Lassen, MD, Principal Investigator — Glostrup Hospital, University of Copenhagen
Locations (1):
- Clinical Trial Unit, Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 subjects were enrolled but 2 subjects were never randomized and have thus not been included in the analysis.
Groups:
- Sangvia and Retransfusion: Blood collected and retransfused with Sangvia.
- Sangvia and no Retransfusion: Blood collected with Sangvia but discarded, i.e. not retransfused.
Period: Overall Study
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Started | 26 | 23
Completed | 26 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14) | 59 (13) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Denmark | 26 | 23 | 49

OUTCOME MEASURES:

1. Secondary Outcome: Plasma Free Hemoglobin (p-Hb) Concentration
Description: Systemic plasma free hemoglobin (p-Hb) concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
g/l
  Screening | 0.2 (0.2) [-0.0288 to 0.1208] | 0.1 (0.1)
  At Randomization (0 hrs) | 0.2 (0.2) | 0.2 (0.2)
  End of transfusion | 1.2 (0.7) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 0.9 (0.7) | 0.1 (0.1)
  6 hours | 0.5 (0.1) | 0.0 (0.1)
  24 hours | 0.1 (0.1) | 0.1 (0.1)
  48 hours | 0.1 (0.1) | 0.1 (0.3)
  96 hours | 0.1 (0.2) | 01. (0.1)

2. Secondary Outcome: Hemoglobin Concentration
Description: Systemic hemoglobin concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
g/dl
  Screening | 14.2 (1.1) | 13.8 (1.3)
  At Randomization (0 hrs) | 11.8 (1.1) | 11.1 (1.5)
  End of transfusion | 12.5 (1.1) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 12.5 (1.1) | 11.6 (1.3)
  6 hours | 12.4 (1.2) | 11.5 (1.2)
  24 hours | 11.6 (1.2) | 10.8 (1.2)
  48 hours | 11.4 (1.0) | 10.8 (1.7)
  96 hours | 11.2 (1.3) | 10.9 (1.5)

3. Secondary Outcome: Potassium Concentration
Description: Systemic potassium concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
mmol/l
  Screening | 4.2 (0.3) | 4.4 (0.4)
  At Randomization (0 hrs) | 4.2 (0.4) | 4.1 (0.7)
  End of transfusion | 4.1 (0.4) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 4.0 (0.4) | 4.3 (0.4)
  6 hours | 4.2 (0.5) | 4.3 (0.4)
  24 hours | 3.9 (0.3) | 4.0 (0.4)
  48 hours | 4.0 (0.6) | 4.0 (0.5)
  96 hours | 4.0 (0.4) | 4.0 (0.5)

4. Secondary Outcome: Creatinine Concentration
Description: Systemic creatinine concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: μmol/l
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
μmol/l
  Screening | 64 (13) | 70 (15)
  At Randomization (0 hrs) | 65 (12) | 69 (16)
  End of transfusion | 68 (13) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 66 (12) | 72 (16)
  6 hours | 62 (12) | 64 (12)
  24 hours | 61 (12) | 66 (17)
  48 hours | 62 (12) | 67 (16)
  96 hours | 59 (12) | 64 (14)

5. Primary Outcome: Difference in Plasma Free Hemoglobin (p-Hb) Concentration
Description: Difference in plasma free hemoglobin (p-Hb) concentration between screening and 24 hours after surgery
Time Frame: At screening and 24 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
g/l | 0.1 (0.2) | 0.0 (0.1)
Statistical Analysis 1: Comparison: Sangvia and Retransfusion vs Sangvia and no Retransfusion; Test type: Non-Inferiority or Equivalence — Information about the size of the standard deviation (SD) for the change was obtained from an earlier study. The SD for the change from pre-operation until 24 hours after start of transfusion was 0.2305. Due to the imprecise measuring device (if values below 0.3 g/l) and the large SD, a non-inferiority margin (∆) of 0.2 g/l was decided to be used in this study, resulting in a total number of 42 evaluable subjects, i.e. 21 subjects per group; p = 0.6294, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Interleukin-1-alpha (IL-1-α) Concentration
Description: Systemic IL-1-α concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 18.36 (24.14) | 23.44 (36.30)
  At Randomization (0 hrs) | 13.66 (18.37) | 22.39 (37.35)
  End of transfusion | 14.97 (16.21) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 14.04 (17.17) | 26.69 (51.07)
  24 hours | 12.45 (14.26) | 22.16 (34.34)
  48 hours | 12.63 (15.06) | 15.74 (14.47)
  96 hours | 13.44 (16.15) | 17.41 (14.10)

7. Secondary Outcome: Interleukin-6 (IL-6) Concentration
Description: Systemic IL-6 concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 8.35 (9.38) | 8.94 (10.45)
  At Randomization (0 hrs) | 7.27 (6.12) | 9.71 (9.71)
  End of transfusion | 37.30 (46.00) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 58.29 (87.34) | 64.20 (93.69)
  24 hours | 116.65 (171.29) | 118.89 (192.73)
  48 hours | 118.05 (163.19) | 163.73 (188.09)
  96 hours | 29.14 (24.00) | 32.51 (19.15)

8. Secondary Outcome: Interleukin-8 (IL-8) Concentration
Description: Systemic IL-8 concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 1.35 (1.07) | 1.35 (0.76)
  At Randomization (0 hrs) | 2.34 (2.67) | 2.01 (2.54)
  End of transfusion | 4.32 (6.41) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 5.17 (9.14) | 2.91 (2.79)
  24 hours | 2.05 (1.53) | 3.13 (2.33)
  48 hours | 2.57 (2.27) | 3.77 (2.88)
  96 hours | 2.48 (1.96) | 2.70 (1.61)

9. Secondary Outcome: Interleukin-10 (IL-10) Concentration
Description: Systemic IL-10 concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 2.25 (2.72) | 2.07 (1.19)
  At Randomization (0 hrs) | 4.59 (3.44) | 7.99 (9.88)
  End of transfusion | 70.65 (100.88) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 50.60 (81.04) | 18.36 (18.11)
  24 hours | 5.29 (4.26) | 4.27 (2.49)
  48 hours | 3.54 (1.48) | 4.96 (3.23)
  96 hours | 2.15 (1.34) | 2.67 (1.12)

10. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-α) Concentration
Description: Systemic TNF-α concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 25.40 (52.70) | 15.42 (34.15)
  At Randomization (0 hrs) | 16.14 (30.51) | 13.87 (28.37)
  End of transfusion | 17.43 (28.41) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 16.23 (28.25) | 14.02 (28.16)
  24 hours | 11.55 (23.60) | 7.86 (17.32)
  48 hours | 9.84 (24.05) | 7.69 (15.98)
  96 hours | 10.37 (20.56) | 5.49 (7.71)

11. Secondary Outcome: Interferon Gamma (IFN-γ) Concentration
Description: Systemic IFN-γ concentration from screening until 96 hours after surgery.
Time Frame: At screening and up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
pg/ml
  Screening | 7.45 (14.17) | 8.61 (18.90)
  At Randomization (0 hrs) | 3.89 (5.35) | 7.37 (15.85)
  End of transfusion | 4.50 (4.24) | NA (NA) — Time point End of transfusion only applicable to subjects in the investigational group (Sangvia and retransfusion).
  3 hours | 4.54 (5.15) | 8.31 (19.15)
  24 hours | 3.94 (3.12) | 7.98 (16.78)
  48 hours | 4.00 (3.49) | 5.94 (7.29)
  96 hours | 4.25 (3.60) | 7.14 (7.18)

12. Secondary Outcome: Mean Blood Loss Volume
Description: Estimated blood loss during and after surgery.
Time Frame: After surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Mean (Full Range); unit: ml
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
ml
  Intra-operative | 623 (444) [150 to 2400] | 742 [200 to 2400]
  Post-operative | 392 [0 to 1150] | 420 [120 to 1525]
  Total | 1015 [150 to 3150] | 1162 [350 to 2800]

13. Secondary Outcome: Frequency of Allogenic Blood Transfusion
Time Frame: Up until 96 hours after surgery (surgery takes place 1-7 days after screening)
Population: All subjects randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Number analyzed (Participants) | 26 | 23
percentage of participants | 8 | 22

ADVERSE EVENTS:
Arm/Group | Sangvia and Retransfusion | Sangvia and no Retransfusion
Serious Adverse Events (participants affected / at risk) | 3/26 | 4/23
Other Adverse Events (participants affected / at risk) | 23/26 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sangvia and Retransfusion (N=26) | Sangvia and no Retransfusion (N=23)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bronchial spasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nerve contusion (Nervous system disorders) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound oozing (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sangvia and Retransfusion (N=26) | Sangvia and no Retransfusion (N=23)
Nausea (Gastrointestinal disorders) | 11 (11) | 6 (6)
Dizziness (Cardiac disorders) | 4 (4) | 5 (5)
Leg pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Hematuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Decreased hemoglobin (Investigations) | 2 (2) | 1 (1)
Fever (General disorders) | 3 (3) | 0 (0)
Syncope (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days